CLINICAL TRIAL: NCT03336775
Title: Efficacy of Acupuncture in Radiotherapy-induced Dysphagia in Patients With Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20160301
Record Dates: First submitted 2016-03-12; First posted 2017-11-08 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Acupuncture
Keywords: acupuncure; dysphagia; radiation
MeSH Terms: conditions — Deglutition Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes, inclduing VDS, rosenbek Penetration-Aspiration Scale scores, opening of upper esophageal sphincter(UES) and excursion of hyoid bone would be evaluated by two radiologists with blind method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Experimental): Patients receive acupuncture for 30 minutes per day for up to 20 sessions (over 4 weeks). These patients also received corticosteroid for 4 weeks, methylprednisolone 80mg ivdrip. for 3 days, 60mg ivdrip. for 3 days, 40mg ivdrip. for 3 days, 30mg po. for 7 days, 20mg po. for 7 days, 10mg po. for 5 days and maintain.
  Interventions: Procedure: acupuncture
- control (No Intervention): Patients receive no acupuncture. The use of corticosteroid is the same with Arm I.

INTERVENTIONS:
Procedure: acupuncture — Acupuncture for 30 minutes per day for up to 20 sessions (over 4 weeks).
  Arms: acupuncture

SUMMARY:
Purpose:

Rationale: Acupuncture is a therapy for physical activity disorders secondary to nervous diseases, and it may have therapeutic effects on dysphagia caused by radiation therapy.

Purpose: This randomized trial aims to investigate whether acupuncture may alleviate radiation-induced dysphagia in patients with head and neck cancer. The effect was compared with outcomes in patients without receiving acupuncture.

DETAILED DESCRIPTION:
OBJECTIVE

Primary:

To determine the therapeutic efficacy of acupuncture on radiotherapy-induced dysphagia in patients with head and neck cancer.

Secondary:

1. To determine whether acupuncture can improve swallow function in these patients.
2. To determine what extent acupuncture can improve the complications of dysphagia of these patients, including the incidence of aspiration pneumonia, malnutrition.
3. To determine what extent this traditional Chinese therapy can improve quality of life of these patients.
4. To evaluate the safety of acupuncture in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive acupuncture for 30 minutes per day for up to 20 sessions (over 4 weeks). These patients also received corticosteroid for 4 weeks, methylprednisolone 80mg ivdrip. for 3 days, 60mg ivdrip. for 3 days, 40mg ivdrip. for 3 days, 30mg po. for 7 days, 20mg po. for 7 days, 10mg po. for 5 days and maintain. Patients undergo VFSS before, at end of therapy (week 4) and 3 months (week 16) after therapy. Swallowing function, outcomes of dysphagia, including incidence of aspiration pneumonia, nutritional status change, and QOL change are assessed at baseline, week 4 and week 16.

Arm Ⅱ: Patients receive corticosteroid only, and the use of corticosteroid is the same with Arm I. Patients undergo VFSS before, at end of therapy (week 4) and 3 months (week 16) after therapy. Swallowing function, outcomes of dysphagia, including incidence of aspiration pneumonia, nutritional status change, and QOL change are assessed at baseline, week 4 and week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received radiation therapy for histologically confirmed head and neck cancer;
2. Prior irradiation >/= 6 months prior to study entry;
3. Age>/= 18 years;
4. Routine laboratory studies with bilirubin </=2 * upper limits of normal (ULN), aspartate aminotransferase (AST or SGOT) < 2 * ULN, creatinine <1.5 * ULN, red-cell count >/= 4,000 per cubic millimeter; white-cell count >/=1500 per cubic millimeter, platelets >/= 75,000 per cubic millimeter; PT, APTT, INR in a normal range;
5. Ability to understand and willingness to sign a written informed consent document, or constant caregivers who well understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Evidence of metastatic disease or tumor recurrence, tumor invasion to major vessels (e.g. the carotid);
2. Evidence of very high intracranial pressure that suggests brain hernia and need surgery;
3. History of seizures or bleeding related to tumor or radiotherapy during or after the completion of radiation;
4. History of coagulation defects or allergy history of contrast agent;
5. History of disorder that affects swallowing, including brain stroke, oral or throat disease, malignances diseases, infection of the nervous system, demyelinating disease, neurodegenerative disease, advanced dementia, diabetes, peripheral vascular disease, HIV infection, familial degenerative peripheral neuropathy;
6. Severe complications: 1) New York heart association grade II or greater congestive heart failure; 2) Serious and inadequately controlled cardiac arrhythmia; 3) Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection); 4) Clinically significant peripheral vascular disease; 5) significant uncontrolled life-threatening infection;
7. Prior use of acupuncture for dysphagia;
8. Enrolled in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The change of Videofluoroscopic Dysphagia Scale (VDS) from baseline to week 4. | Assessed at baseline and week 4 during acupuncture treatment.
  The change of Videofluoroscopic Dysphagia Scale (VDS) from baseline to week 4. VDS, according to result of Video Fluoroscopy Swallowing Study (VFSS), used as an objective and quantifiable predictor of recovery of the swallowing function. A videofluoroscopic dysphagia scale (VDS) with a sum of 100 was made according to the odds ratios of prognostic factors. The validity of the scale was evaluated by using a receiver operating characteristic curve. The VDS was compiled using the following 14 items: lip closure, bolus formation, mastication, apraxia, tongue-to-palate contact, premature bolus loss, oral transit time, triggering of pharyngeal swallow, vallecular residue, laryngeal elevation, pyriform sinus residue, coating of pharyngeal wall, pharyngeal transit time, and aspiration. At a scale cutoff value of 47. The higher the VDS score, the worse the swallowing function.

SECONDARY OUTCOMES:
The change of Videofluoroscopic Dysphagia Scale (VDS) from baseline to week 16. | Assessed at baseline and 12 weeks post acupuncture treatment.
  The change of Videofluoroscopic Dysphagia Scale (VDS) from baseline to week 16. VDS, according to result of Video Fluoroscopy Swallowing Study (VFSS), used as an objective and quantifiable predictor of recovery of the swallowing function. A videofluoroscopic dysphagia scale (VDS) with a sum of 100 was made according to the odds ratios of prognostic factors. The validity of the scale was evaluated by using a receiver operating characteristic curve. The VDS was compiled using the following 14 items: lip closure, bolus formation, mastication, apraxia, tongue-to-palate contact, premature bolus loss, oral transit time, triggering of pharyngeal swallow, vallecular residue, laryngeal elevation, pyriform sinus residue, coating of pharyngeal wall, pharyngeal transit time, and aspiration. At a scale cutoff value of 47. The higher the VDS score, the worse the swallowing function.
The change of rosenbek Penetration-Aspiration Scale scores, opening of upper esophageal sphincter(UES) and excursion of hyoid bone from baseline to week 4 and week 16. | Assessed at baseline, week 4 during acupuncture treatment and 12 weeks post acupuncture treatment.
  The rosenbek Penetration-Aspiration Scale(PAS) scores, opening of upper esophageal sphincter(UES) and excursion of hyoid bone will be assessed according to the VFSS to objectively evaluate the swallowing function. Penetration deﬁned as passage of the bolus content into the laryngeal vestibule above the vocal cords. When food crossed the vocal cords and entered the airways, it was considered aspiration. Records were taken of the moment aspiration occurred (before onset of pharyngeal swallow, during pharyngeal contraction, or after swallowing). Consideration was also given to the appearance or not of cough during aspiration. Silent aspiration was deﬁned as the entry of food below the level of the true vocal cords, without cough or any outward sign of difﬁculty. The PAS score with a total of 8, and >2 is considered to be abnormal. The higher the PAS score, the worse the swallowing function.
The incidence of aspiration pneumonia change from baseline to week 4 and week 16. | Assessed at baseline, week 4 during acupuncture treatment and 12 weeks post acupuncture treatment.
  The incidence of aspiration pneumonia change from baseline to week 4 and week 16.
The change of nutritional status from baseline to week 4 and week 16. | Assessed at baseline, week 4 during acupuncture treatment and 12 weeks post acupuncture treatment.
  The change of nutritional status from baseline to week 4 and week 16. The nutritioanl status include the weight, BMI, albumin.
The percentage of necessary of nasogastric feeding and gastrostomy from baseline to week 16. | Assessed at baseline and 12 weeks post acupuncture treatment.
  The percentage of necessary of nasogastric feeding and gastrostomy from baseline to week 16.
The change of Quality of Life (QOL) scores from baseline to week 4 and week 16. | Assessed at baseline, week 4 during acupuncture treatment and 12 weeks post acupuncture treatment.
  The change of Quality of Life (QOL) scores from baseline to week 4 and week 16. The WHOQOL-BREF instrument comprises 26 items, which measures the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF (Field Trial Version) produces a quality of life profile. It is possible to derive four domain scores. The four domain scores denote an individual's perception of quality of life in each particular domain. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100.

CONTACTS AND LOCATIONS:
Overall Officials: yamei tang, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No